CLINICAL TRIAL: NCT03774810
Title: Three Approaches to Maintenance Therapy for Chronic Insomnia in Older Adults
Brief Title: Partial Reinforcement II: Three Approaches to Maintenance Therapy for Chronic Insomnia
Acronym: R01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 831801; R01AG054521-01A1 (NIH)
Record Dates: First submitted 2018-12-10; First posted 2018-12-13 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Insomnia; Insomnia Chronic
Keywords: insomnia; sleep; chronic insomnia; zolpidem; ambien
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Continuous (Experimental): Nightly active dose (QHS). The intervention is zolpidem tartrate 5 mg or 10 mg.
  Interventions: Drug: Zolpidem tartrate
- Partial Reinforcement 1 (Experimental): 1 active dose per week with 6 placebos interspersed between the active dose. The intervention is zolpidem tartrate 5 mg or 10 mg.
  Interventions: Drug: Zolpidem tartrate
- Partial Reinforcement 3 (Experimental): 3 active doses per week with 4 placebos interspersed between the active doses. The intervention is zolpidem tartrate 5 mg or 10 mg.
  Interventions: Drug: Zolpidem tartrate
- Low Frequency Intermittent Dosing (Experimental): 1 to 3 active doses per week, on night chosen by participant (as needed). The intervention is zolpidem tartrate 5 mg or 10 mg.
  Interventions: Drug: Zolpidem tartrate

INTERVENTIONS:
Drug: Zolpidem tartrate — Zolpidem Tartrate, 5mg for men older than 60 and women of all ages. 10 mg for men younger than 60.
  Other Names: zolpidem; ambien

SUMMARY:
The study is a three phase sequential study of the medical treatment of insomnia with zolpidem. All participating subjects will receive one month of standard nightly treatment. If the subject has a positive treatment response they continue in the study and are randomized to one of four conditions: intermittent dosing (3-5 pills week, full dose), or one of three variable dose conditions (nightly pill use where any given pill is a variable dose). Standard treatment will last for 4 weeks. The experimental phase will extend over two periods. The first period will last for 12 weeks. The second period will last for 36 weeks. Both periods include:

• Taking a pill 30 minutes prior to bedtime.

In one case, this will involve taking 3-5 pills per week. In the remaining condition pills will be taken on each and every night. Depending on the specific group that the subject is assigned to, they will either receive 10mg or 5mg of zolpidem (variable by age and sex) or a variable dose of zolpidem on a nightly basis (range from 0 mg to 10 mg per night).

* Completing a sleep diary each day;
* Completing 6 to 7 questionnaires each week;
* A monthly visit to Penn to return your medication foil packs and to receive a new foil pack with the next month of medication.

During Phases 3&4, the subject will be asked to undergo quarter annual physicals so that we can optimally track their health and wellbeing. The physicals will involve standard vitals measures (e.g., temperature, blood pressure, height and weight, etc.) and, based on the judgement of the research clinician, may involve an EKG and blood and urine chemistries.

If the subject does not experience a treatment response or (following a treatment response) experiences a relapse of insomnia, they will not continue in the study but will be given the opportunity to be treated with Cognitive Behavioral Therapy for Insomnia (CBT-I) at no cost. Assessments of the subjects clinical status will be based on your daily sleep diaries and weekly questionnaires.

DETAILED DESCRIPTION:
Phase-1: Initial Evaluation.

This evaluation occurs at the offices of the Behavioral Sleep Medicine Program (Suite 670, 3535 Market Street Philadelphia, PA 19104) and lasts about 1 to 2 hours. Procedures include:

* Completing forms asking questions about your sleep, mood, alcohol use, medical history, your current medications, and background questions about your age, race, and education.
* The provision of your consent to contact your primary care provider to gain their assent (agreement) that you may participate in the trial safely.

The information obtained during the initial assessment will be used to see if you are eligible to participate in this study. If you are determined ineligible, you will not be able to continue in the study but will be provided with a referral if appropriate.

NOTE: This study will be using an Internet Data Portal (IDP) system to collect most questionnaire data. The IDP is a Research Electronic Data Capture and is a secure web application. It is a password protected site located on Penn's servers in which the data will live in a database online where only qualified research personnel can access it. During the initial evaluation you will be introduced to this system and provided with a username and password. The study staff will assist you in filling out the questionnaires using this IDP system.

Phase-2: Baseline Period.

This phase lasts 14 days. Your participation includes:

* Completing daily sleep diaries at home. The online diary form requires about 5 minutes each day to complete.
* Completing 6 to 7 forms asking questions about your medical symptoms, and sleep each week of the baseline period. These online questionnaires require about 15 minutes to complete.
* Abstaining from the use of any medication or over the counter product that is used expressly for the purpose of helping you fall or stay asleep (e.g. trazadone/Desyrel, melatonin, Nyquil, Tylenol PM, Benadryl, etc.). If you choose to discontinue your current sleep medication to participate in our study, please do this in consultation with the clinician that prescribed your sleep medication. Please note that discontinuation of your current sleep medication will make it necessary to extend the baseline component of our study by at least two weeks. Should the sleep diaries indicate that your insomnia is not of the type, severity, or frequency required for the study, you will not be able to continue in the study but will be provided with a referral. This referral will be for the Penn Sleep Disorder Center. If you or study personnel deem your two weeks to be unusual, you may be offered the chance to repeat the baseline period.

Phase-3: Sleep Lab Study (polysomnography) or Home Sleep Apnea Test (HSAT). You will undergo a polysomnography study or an HSAT to determine if you are eligible to continue in the study. During the pandemic all sleep tests will be administered at home. After the pandemic, the study investigators will decide which type of study you will receive. Both sleep assessments will last for 1 night.

The HSAT equipment will be shipped to your house. A member of the study team will contact you to go over proper use instructions. On the night of the test, you can go to bed at your regular bedtime. Prior to bedtime, you will attach the sensor(s) as instructed and start the test. Upon waking up, you will stop the test and remove the sensor(s). On the day immediately following the sleep test, you will ship the device back in the prepaid shipping envelope Procedures for the polysomnography study are: you will be asked to arrive at the sleep lab located at the Hospital of the University of Pennsylvania (HUP) at the cross streets of 34th and Spruce by 7 P.M. for a polysomnographic study (PSG). Upon arrival, to ensure for accurate laboratory measurements, urine toxicology screens may be performed to rule out illegal substance use. These data are acquired to explain abnormal findings on the PSG. Following the sleep study, it will be determined whether a repeat study is necessary based on the findings both from the clinical chemistries and the polysomnography. If a repeat study is necessary, one of the project investigators will discuss the issue of substance use with you to: (1) determine if the clinical chemistries' finding was an error (for example poppy seeds led to a positive screen) or (2) gain your willingness to refrain from substance use for the second PSG and for the remainder of the study. If you screen positive a second time, your participation will be discontinued.

The specific procedure for a PSG requires that you have a set of sensors placed on your face, scalp, and body by a technician. All the sensors are attached with surgical tape, paste and glue. The sensors on your face are attached on your left and right temple, cheek bone and under your nose. The sensors on the temple and cheek bone measure eye movements associated with falling asleep and dreaming. The sensors under your nose measure airflow through your mouth and nose. The sensors on your scalp measure brain waves during sleep. The sensors on the body are placed above the collar bones and over the calf muscles. The sensors over the collar bones measure heart muscle activity. The sensors over the calf muscles measure muscle activity from the legs. In addition, a strap will be placed around your chest and abdomen to measure respiration.

After you have been connected to the equipment, you are expected to stay in bed until final wake time the next morning, except for bathroom breaks. You will be visually monitored by the lab technicians by remote video. In the morning, you will be awakened by the technician (if needed), be unhooked from the equipment, and then allowed to shower, dress, and eat before leaving. You will be free to go about your normal schedule for the rest of the day.

If the in-lab PSG sleep or HSAT study finds evidence of a sleep disorder other than insomnia, such as sleep apnea, you will not be able to continue in the study but will be provided with a referral.

Phase-4: Standard Treatment. All participating subjects will receive one month of standard nightly treatment. If you have a positive treatment response you will remain in the study and be randomized to one of the following treatment conditions: nightly dosing, intermittent dosing (1-3 pills week, full dose), or one of two variable dose conditions (nightly pill use where any given pill is a variable dose). The assignment of condition will be accomplished by a process that is the same as the flip of a coin and neither you nor the study personnel will know which condition you have been assigned to (this is referred to as a "double blind" study). You will have an equal chance of being randomized to each of the 4 study arms. In the case of an emergency, the blind will be broken and the study doctor and clinicians associated with your care will be informed of which dosing condition you were assigned to.

Standard treatment will last for 4 weeks. The experimental phase will extend over two periods. The first period will last for 12 weeks. The second period will last for 36 weeks.

Both periods include:

* Taking a pill 30 minutes prior to bedtime. In one case, this will involve taking 1-3 pills per week. In the remaining conditions, pills will be taken on each and every night. Depending on the specific group you are assigned to, you will either receive 10mg or 5mg of zolpidem (variable by age and sex) or a variable dose of zolpidem on a nightly basis (range from 0 mg to 10 mg per night). Please note that the effect of zolpidem may be slowed if taken with or immediately after a meal.
* Completing a sleep diary each day;
* Completing 6 to 7 questionnaires each week;
* A monthly visit to Penn to return your medication foil packs and to receive a new foil pack with the next month of medication.

If you do not experience a treatment response or (following a treatment response) you experience a relapse of insomnia, you will not be able to continue in the study but will be given the opportunity to be treated with Cognitive Behavioral Therapy for Insomnia (CBT-I) at no cost. Assessments of your clinical status (how your insomnia is responding to treatment) will be based on your daily sleep diaries and weekly questionnaires.

During Phase-4, you will be asked to undergo quarter annual physicals so that we can optimally track your health and wellbeing. The physicals will involve standard vital measures (e.g., temperature, blood pressure, height and weight, etc.) and, based on the judgement of the research clinician, may involve an EKG and/or blood and urine chemistries.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for Insomnia Disorder, ICSD-3, and RDC criteria for Psychophysiologic Insomnia
* Age 40-85

Exclusion Criteria:

* currently in treatment for insomnia
* unstable medical or psychiatric illness
* a history of treatment failure with zolpidem
* discontinuation of zolpidem owing to side effects
* current experience, or history, of parasomnias (within the last 5 years)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Perlis, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here to learn about our available studies — http://www.sleeplessinphilly.com
- See also: Click here to learn more about our sleep research laboratory — http://www.med.upenn.edu/bsm/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 197 subjects were consented and enrolled into baseline.
Pre-assignment Details: 7 subjects were lost to follow-up.
  13 subjects withdrew during baseline.
  28 did not meet criteria for Insomnia based on baseline sleep diaries.
  34 were screened out for sleep apnea.
  115 continued to phase 1 of treatment
Groups:
- QHS-FD (Phase 1); Full Dose Nightly (QHS-FD) (Phases 2 & 3): Nightly active dose (QHS). The intervention is zolpidem tartrate 5 mg or 10 mg.
  Zolpidem tartrate: Zolpidem Tartrate, 5mg for men 60 and older and women of all ages. 10 mg for men younger than 60.
- Partial Reinforcement 1 (PR1) (Phases 2 & 3): 1 active dose per week with 6 placebos interspersed between the active dose. The intervention is zolpidem tartrate 5 mg or 10 mg.
  Zolpidem tartrate: Zolpidem Tartrate, 5mg for men 60 and older and women of all ages. 10 mg for men younger than 60.
- Partial Reinforcement 3 (PR3) (Phases 2 & 3): 3 active doses per week with 4 placebos interspersed between the active doses. The intervention is zolpidem tartrate 5 mg or 10 mg.
  Zolpidem tartrate: Zolpidem Tartrate, 5mg for men 60 and older and women of all ages. 10 mg for men younger than 60.
- Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3): 1 to 3 active doses per week, on night chosen by participant (as needed). The intervention is zolpidem tartrate 5 mg or 10 mg.
  Zolpidem tartrate: Zolpidem Tartrate, 5mg for men 60 and older and women of all ages. 10 mg for men younger than 60.
Period: Phase 1
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Started | 115 | 0 | 0 | 0 | 0
Completed | 83 | 0 | 0 | 0 | 0
Not Completed | 32 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 21 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0
Period: Phase 2 (3 Months)
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Started | 0 | 22 | 18 | 23 | 20
Completed | 0 | 13 | 14 | 17 | 18
Not Completed | 0 | 9 | 4 | 6 | 2
Not completed — Lack of Efficacy | 0 | 3 | 2 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 2 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Period: Phase 3 (9-month Extension of Phase 2)
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Started | 0 | 13 | 14 | 17 | 18
Completed | 0 | 9 | 9 | 10 | 12
Not Completed | 0 | 4 | 5 | 7 | 6
Not completed — Lack of Efficacy | 0 | 3 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 5 | 2
Not completed — Withdrawn by PI due to study end. | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All subjects received the same treatment for phase 1, so none were randomized to other conditions.
Groups:
- QHS-FD (Phase 1): 1 to 3 active doses per week, on night chosen by participant (as needed). The intervention is zolpidem tartrate 5 mg or 10 mg.
  Zolpidem tartrate: Zolpidem Tartrate, 5mg for men 60 and older and women of all ages. 10 mg for men younger than 60.
- Partial Reinforcement 1 (PR1) (Phases 2 & 3): 1 active doses/week with 6 placebos interspersed between active doses.
  Active Doses: zolpidem tartrate 5 mg (males 60+ years of age, all females) or 10 mg (males 40-59 years of age).
- Partial Reinforcement 3 (PR3) (Phases 2 & 3): 3 active doses/week with 4 placebos interspersed between active doses.
  Active Doses: zolpidem tartrate 5 mg (males 60+ years of age, all females) or 10 mg (males 40-59 years of age).
- Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3): 1-3 active doses per week, on night(s) chosen by participant (as needed).
  Active Doses: zolpidem tartrate 5 mg (males 60+ years of age, all females) or 10 mg (males 40-59 years of age).
- Full Dose Nightly (QHS-FD) (Phases 2 & 3): Nightly active dose (QHS).
  Active Doses: zolpidem tartrate 5 mg (males 60+ years of age, all females) or 10 mg (males 40-59 years of age).
- Total: Total of all reporting groups
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3) | Total
Number analyzed (Participants) | 115 | 0 | 0 | 0 | 0 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (8.3) |  |  |  |  | 56.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 0 | 0 | 0 | 0 | 87
  Male | 28 | 0 | 0 | 0 | 0 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 113 | 0 | 0 | 0 | 0 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 0 | 0 | 0 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 0 | 0 | 0 | 0 | 6
  White | 100 | 0 | 0 | 0 | 0 | 100
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 115 |  |  |  |  | 115
Sleep Continuity [Mean (Standard Deviation); unit: Minutes] — Average baseline sleep diary sleep continuity variables
  Minutes
    Sleep Latency | 31.71 (42.98) |  |  |  |  | 31.71 (42.98)
    Wake After Sleep Onset | 50.54 (50.54) |  |  |  |  | 50.54 (47.67)
    Early Morning Awakenings | 74.9 (56.84) |  |  |  |  | 74.79 (56.84)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response (Phase 1)
Description: Tracking treatment response via assessing daily sleep continuity (sleep latency, wake after sleep onset, and early morning awakenings).
Time Frame: 1 Month
Population: All subjects received the same treatment for phase 1, so none were randomized to other conditions.
Measure: Count of Participants; unit: Participants
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Number analyzed (Participants) | 115 | 0 | 0 | 0 | 0
Participants | 94 |  |  |  |

2. Primary Outcome: Insomnia Relapse (Phase 2)
Description: Tracking relapse via assessing daily sleep continuity (sleep latency, wake after sleep onset, and early morning awakenings).
Time Frame: 3 months
Population: This outcome only includes phase 2, so, by definition the phase 1 group had no subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Number analyzed (Participants) | 0 | 22 | 18 | 23 | 20
Participants |  | 4 | 3 | 3 | 1

3. Secondary Outcome: Sleep Continuity (Phase 1)
Description: Assess sleep continuity by assessing daily sleep diary responses.
Time Frame: 1 Month
Population: This outcome only includes phase 1, so, by definition the groups for phases 2 and 3 had no subjects.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Number analyzed (Participants) | 115 | 0 | 0 | 0 | 0
Minutes
  Sleep Latency (SL) | 17.35 (26.09) |  |  |  |
  Wake After Sleep Onset (WASO) | 29.46 (34.82) |  |  |  |
  Early Morning Awakenings (EMA) | 69.07 (52.45) |  |  |  |

4. Secondary Outcome: Sleep Continuity (Phase 2)
Description: Assess sleep continuity by assessing daily sleep diary responses.
Time Frame: 3 months
Population: This outcome only includes phase 2, so, by definition the phase 1 group had no subjects.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Number analyzed (Participants) | 0 | 22 | 18 | 23 | 20
Minutes
  Sleep Latency (SL) |  | 21.24 (26.51) | 24.56 (45.02) | 21.76 (31.38) | 13.03 (20.37)
  Wake After Sleep Onset (WASO) |  | 37.51 (39.07) | 44.29 (50.74) | 34.20 (38.31) | 22.78 (28.46)
  Early Morning Awakenings (EMA) |  | 64.77 (51.79) | 69.88 (57.33) | 65.61 (52.56) | 53.52 (36.06)

5. Secondary Outcome: Sleep Continuity (Phase 3)
Description: Assess sleep continuity by assessing daily sleep diary responses.
Time Frame: 9 months
Population: This outcome only includes phase 3, so, by definition the phase 1 group had no subjects.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Number analyzed (Participants) | 0 | 13 | 14 | 17 | 18
Minutes
  Sleep Latency (SL) |  | 20.32 (27.51) | 29.71 (52.42) | 24.32 (35.00) | 11.43 (14.09)
  Wake After Sleep Onset (WASO) |  | 34.73 (38.33) | 38.10 (42.09) | 37.80 (41.00) | 21.25 (28.10)
  Early Morning Awakenings (EMA) |  | 59.34 (44.21) | 79.12 (68.48) | 62.68 (48.73) | 50.19 (36.49)

6. Primary Outcome: Insomnia Relapse (Phase 3)
Description: as for outcome 2
Time Frame: 9 months
Population: This outcome only includes phase 3, so, by definition the phase 1 group had no subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
Number analyzed (Participants) | 0 | 13 | 14 | 17 | 18
Participants |  | 3 | 3 | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 13 months per subject.
Description: No serious adverse events occurred.
Groups:
- Full Dose Nightly (QHS-FD) (Phases 2 & 3): Nightly active dose (QHS). The intervention is zolpidem tartrate 5 mg or 10 mg.
  Zolpidem tartrate: Zolpidem Tartrate, 5mg for men older than 60 and women of all ages. 10 mg for men younger than 60.
Arm/Group | QHS-FD (Phase 1) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) | Full Dose Nightly (QHS-FD) (Phases 2 & 3)
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/22 | 0/18 | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/22 | 0/18 | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 2/115 | 4/22 | 7/18 | 2/23 | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QHS-FD (Phase 1) (N=115) | Partial Reinforcement 1 (PR1) (Phases 2 & 3) (N=22) | Partial Reinforcement 3 (PR3) (Phases 2 & 3) (N=18) | Low Frequency Intermittent Dosing (IDS-FD) (Phases 2 & 3) (N=23) | Full Dose Nightly (QHS-FD) (Phases 2 & 3) (N=20)
Brain Fog (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Daytime Sleepiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Scotomas (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Torn anterior cruciate ligament (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Jitteriness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypnic Jerks (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach Aches/Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic Attacks (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Worsening Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phantosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The following results are preliminary and do not take into account post-randomization factors such as missing data, dropout, or adherence to the intervention regimens. Accordingly, the results are considered preliminary and will be updated on or before the new year (2025).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03774810/Prot_SAP_005.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03774810/ICF_001.pdf